CLINICAL TRIAL: NCT00458900
Title: Pharmacokinetic Evaluation of Moxifloxacin IV to Enteral Switch Therapy in Intensive Care Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007/071
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IV and enteral administration of moxifloxacin (Experimental): IV and enteral administration of moxifloxacin
  Interventions: Drug: IV and enteral administration of moxifloxacin

INTERVENTIONS:
Drug: IV and enteral administration of moxifloxacin — IV and enteral administration of moxifloxacin

SUMMARY:
In the Intensive Care (IC)-unit moxifloxacin treatment is often started with intravenous administrations. As moxifloxacin is known to have a high oral bioavailability in healthy volunteers, patients are switched to oral or enteral therapy as soon as possible. However, no data on plasma levels for moxifloxacin during such a switch-therapy in IC-patients are available. Therefore, this study aims to evaluate the moxifloxacin-plasma levels and their inter-individual variability during IV to enteral switch therapy in IC-patients.

ELIGIBILITY:
Inclusion Criteria:

* IC patients treated with 400 mg moxifloxacin IV (once a day) that can be switched to enteral administration of 400 mg moxifloxacin.
* IV steady state
* Hemodynamic stability
* Normal enteral feeding without prokinetics
* Presence of arterial line
* Informed consent
* ≥ 18 jaar

Exclusion Criteria:

* Dialysis patients
* Creatinine clearance < 30 ml/min
* Transaminase levels > 5x upper limit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 2 days
  Pharmacokinetics will be followed.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Colpaert, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be